CLINICAL TRIAL: NCT02205333
Title: A Phase 1b/2, Open-label Study to Evaluate the Safety and Tolerability of MEDI6469 in Combination With Immune Therapeutic Agents or Therapeutic Monoclonal Antibodies in Subjects With Selected Advanced Solid Tumors or Aggressive B-cell Lymphomas
Brief Title: A Phase 1b/2 Safety and Tolerability Study of MEDI6469 in Combination With Therapeutic Immune Agents or Monoclonal Antibodies
Acronym: MEDI6469
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early at the sponsor's discretion.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4981C00001
Record Dates: First submitted 2014-07-18; First posted 2014-07-31 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Advanced Solid Tumors; Aggressive B-cell Lymphomas
Keywords: Advanced Solid tumors; Diffuse Large B-cell Lymphoma; programmed death 1; programmed dealth ligand 1; cytotoxic T-lymphocyte-associated antigen-4; OX40 ligand
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tremelimumab; durvalumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- MEDI6469 6 mg/kg (Experimental): Participants received MEDI6469 6 milligram/kilogram (mg/kg) as a single intravenous (IV) administration on Day 1
  Interventions: Biological: MEDI6469 Monotherapy
- MEDI6469 10 mg/kg (Experimental): Participants received MEDI6469 10 mg/kg as a single IV administration on Day 1
  Interventions: Biological: MEDI6469 Monotherapy
- MEDI6469 2 mg/kg+Tremelimumab 3 mg/k (Experimental): Participants received MEDI6469 2 mg/kg as a single IV administration on Day 1 plus tremelimumab 3 mg/kg as IV administration on Day 1 then every 4 weeks (Q4W) for 6 doses, after which every 12 weeks (Q12W) for 2 doses or until PD
  Interventions: Biological: MEDI6469 Plus Tremelimumab
- MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg (Experimental): Participants received MEDI6469 2 mg/kg as a single IV administration on Day 1 plus tremelimumab 10 mg/kg as IV administration on Day 1 then Q4W for 6 doses after which Q12W for 2 doses or until progression of disease (PD)
  Interventions: Biological: MEDI6469 Plus Tremelimumab
- MEDI6469 2 mg/kg+Durvalumab 3 mg/kg (Experimental): Participants received MEDI6469 2 mg/kg as a single IV administration on Day 1 plus durvalumab 3 mg/kg as IV administration on Day 1 then every 2 weeks (Q2W) for 12 months or until PD
  Interventions: Biological: MEDI6469 Plus Durvalumab
- MEDI6469 2 mg/kg+Durvalumab 10 mg/kg (Experimental): Participants received MEDI6469 2 mg/kg as a single IV administration on Day 1 plus durvalumab 10 mg/kg as IV administration on Day 1, then Q2W for 12 months or until PD
  Interventions: Biological: MEDI6469 Plus Durvalumab
- MEDI6469 10 mg/kg+Durvalumab 10 mg/kg (Experimental): Participants received MEDI6469 10 mg/kg as a single IV administration on Day 1 plus durvalumab 10 mg/kg as IV administration on Day 1, then Q2W for 12 months or until PD
  Interventions: Biological: MEDI6469 Plus Durvalumab
- MEDI6469 2 mg/kg+Rituximab 375 mg/m^2 (Experimental): Participants received MEDI6469 2 mg/kg as a repeat IV administration on Day 3 then Q4W for 11 doses, or until confirmed complete response (CR) plus 1 cycle, or PD plus rituximab 375 mg/m^2 as IV administration on Days 1, 8, and 29; then Q4W for 10 doses, or until confirmed CR plus 1 cycle, or PD
  Interventions: Biological: MEDI6469 plus Rituximab
- MEDI6469 10 mg/kg+Rituximab 375 mg/m^2 (Experimental): Participants received MEDI6469 10 mg/kg as a repeat IV administration on Day 3 then Q4W for 11 doses, or until confirmed CR plus 1 cycle, or PD plus rituximab 375 mg/m2 as IV administration on Days 1, 8, and 29; then Q4W for 10 doses, or until confirmed CR plus 1 cycle, or PD
  Interventions: Biological: MEDI6469 plus Rituximab

INTERVENTIONS:
Biological: MEDI6469 Monotherapy — single intravenous (IV) administration of MEDI6469
  Arms: MEDI6469 10 mg/kg; MEDI6469 6 mg/kg
Biological: MEDI6469 Plus Tremelimumab — MEDI6469 in combination with Tremelimumab
  Arms: MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg; MEDI6469 2 mg/kg+Tremelimumab 3 mg/k
Biological: MEDI6469 Plus Durvalumab — MEDI6469 in combination with Durvalumab
  Arms: MEDI6469 10 mg/kg+Durvalumab 10 mg/kg; MEDI6469 2 mg/kg+Durvalumab 10 mg/kg; MEDI6469 2 mg/kg+Durvalumab 3 mg/kg
Biological: MEDI6469 plus Rituximab — MEDI6469 in combination with Rituximab
  Arms: MEDI6469 10 mg/kg+Rituximab 375 mg/m^2; MEDI6469 2 mg/kg+Rituximab 375 mg/m^2

SUMMARY:
The main purpose of this study is to determine the best dose of MEDI6469 that is safe and tolerable when given as monotherapy and in combination with tremelimumab, MEDI4736 (durvalumab), or rituximab in participants with either advanced solid tumors or diffuse large B-cell lymphoma (DLBCL). Tremelimumab and MEDI4736 (durvalumab) will be tested with MEDI6469 in a set of participants with advanced solid tumors while rituximab will be tested with MEDI6469 in participants with DLBCL. MEDI6469 will be tested as monotherapy in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adults >/= 18 years old
* Histologically or cytologically confirmed advanced solid tumors that are refractory to standard therapy or for which no standard therapy exists (Monotherapy and in Cohorts A and B)
* At least one lesion measurable by RECIST not previously irradiated (Monotherapy and in Cohorts A and B)
* Histologically confirmed DLBCL(Cohort C)
* Adequate organ and marrow function
* ECOG performance status of 0 or 1
* Willingness to provide consent for biopsy samples

Exclusion Criteria:

* Prior exposure to immunotherapy (either as a single agent or in combination) including but not limited to CD137 or OX40 agonists, anti-CTLA-4, anti-PD-1, or anti-PD-L1, anti-PD-L2 antibody or pathway-targeting agents
* History of organ transplant that requires use of immunosuppressives
* History of primary immunodeficiency or tuberculosis
* Active or prior documented autoimmune disease within the past 3 years
* Active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months
* Major surgical procedure within 30 days prior to the first dose of investigational product or still recovering from prior surgery
* Women who are pregnant or lactating

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune, LLC, Study Director — MedImmune LLC
Locations (13):
- United States (13):
  - Research Site, Scottsdale, Arizona
  - Research Site, Sacramento, California
  - Research Site, Santa Monica, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Detroit, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Hackensack, New Jersey
  - Research Site, Huntersville, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 58 participants were screened at 13 sites in the United States of America (USA).
Pre-assignment Details: A total of 58 participants were screened for this study, of which 48 participants were enrolled and received study treatment.
Groups:
- MEDI6469 6 Milligram/Kilogram (mg/kg): Participants received MEDI6469 6 mg/kg as a single intravenous (IV) administration on Day 1
- MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg: Participants received MEDI6469 2 mg/kg as a single IV administration on Day 1 plus tremelimumab 3 mg/kg as IV administration on Day 1, then every 4 weeks (Q4W) for 6 doses, after which every 12 weeks (Q12W) for 2 doses or until PD
- MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg: Participants received MEDI6469 2 mg/kg as a single IV administration on Day 1 plus tremelimumab 10 mg/kg as IV administration on Day 1, then Q4W for 6 doses, after which Q12W for 2 doses or until PD
- MEDI6469 2 mg/kg+Durvalumab 3 mg/kg: Participants received MEDI6469 2 mg/kg as a single IV administration on Day 1 plus durvalumab 3 mg/kg as IV administration on Day 1, then every 2 weeks (Q2W) for 12 months or until PD
- MEDI6469 2 mg/kg+Rituximab 375 mg/m^2: Participants received MEDI6469 2 mg/kg as a repeat IV administration on Day 3 then Q4W for 11 doses, or until confirmed complete response (CR) plus 1 cycle or PD plus rituximab 375 mg/m^2 as IV administration on Days 1, 8, and 29; then Q4W for 10 doses, or until confirmed CR plus 1 cycle, or PD
- MEDI6469 10 mg/kg+Rituximab 375 mg/m^2: Participants received MEDI6469 10 mg/kg as a repeat IV administration on Day 3, then Q4W for 11 doses, or until confirmed CR plus 1 cycle, or PD plus rituximab 375 mg/m^2 as IV administration on Days 1, 8, and 29; then Q4W for 10 doses, or until confirmed CR plus 1 cycle, or PD
Period: Overall Study
Arm/Group | MEDI6469 6 Milligram/Kilogram (mg/kg) | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg+Rituximab 375 mg/m^2
Started | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Completed | 2 | 0 | 1 | 0 | 1 | 4 | 2 | 1 | 1
Not Completed | 6 | 6 | 2 | 7 | 5 | 3 | 5 | 2 | 0
Not completed — Death | 5 | 6 | 2 | 6 | 5 | 3 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI6469 6 Milligram/Kilogram (mg/kg) | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg+Rituximab 375 mg/m^2 | Total
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (12.6) | 63.8 (8.9) | 48.0 (6.9) | 61.3 (8.7) | 57.5 (19.4) | 66.6 (14.5) | 62.6 (9.1) | 70.3 (4.6) | 73.0 (NA) — Not evaluable due to insufficient number of participants. | 61.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 2 | 3 | 1 | 3 | 1 | 0 | 20
  Male | 3 | 3 | 1 | 5 | 3 | 6 | 4 | 2 | 1 | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of MEDI6469
Description: The MTD was the highest dose within a cohort where no more than 1 out of 6 participants experienced dose-limiting toxicities (DLTs) or the highest protocol-defined dose for each agent in the absence of exceeding the MTD.
Time Frame: From the first dose of study treatment through 28 days after the first dose (up to 28 days)
Population: DLT-evaluable population: All participants enrolled in the dose-escalation phase who received study treatment per protocol during the first 28 days and completed safety follow-up through the DLT-evaluation period or experienced any DLT.
Measure: Number; unit: milligram per kilogram (mg/kg)
Groups:
- MEDI6469 6 mg/kg: Participants received MEDI6469 6 mg/kg as a single intravenous (IV) administration on Day 1
- MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2: Participants received MEDI6469 2 mg/kg as a repeat IV administration on Day 3 then Q4W for 11 doses or until confirmed complete response (CR) plus 1 cycle or PD plus rituximab 375 mg/m^2 as IV administration on Days 1, 8, and 29; then Q4W for 10 doses, or until confirmed CR plus 1 cycle, or PD
- MEDI6469 10 mg/kg + Rituximab 375 mg/m^2: Participants received MEDI6469 10 mg/kg as a repeat IV administration on Day 3, then Q4W for 11 doses, or until confirmed CR plus 1 cycle, or PD plus rituximab 375 mg/m^2 as IV administration on Days 1, 8, and 29; then Q4W for 10 doses, or until confirmed CR plus 1 cycle, or PD
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
milligram per kilogram (mg/kg) | NA — Dose escalation was completed without determination of MTD. | NA — Dose escalation was completed without determination of MTD. | NA — Dose escalation was terminated early prior to completion of the protocol-specified dose ranges. | NA — Dose escalation was terminated early prior to completion of the protocol-specified dose ranges. | NA — Dose escalation was completed without determination of MTD. | NA — Dose escalation was completed without determination of MTD. | NA — Dose escalation was completed without determination of MTD. | NA — Dose escalation was terminated early prior to completion of the protocol-specified dose ranges. | NA — Dose escalation was terminated early prior to completion of the protocol-specified dose ranges.

2. Primary Outcome: Number of Participants With DLTs
Description: The DLT was any Grade 3 or higher treatment-related toxicity (including liver transaminase elevation higher than 8×upper limit of normal [ULN] or total bilirubin higher than 5×ULN; any >=Grade 2 pneumonitis that did not resolve to <=Grade 1 within 3 days) that occurred during the DLT time frame, and excluded the following: Grade 3 fatigue for less than or equal to (<=) 7 days; Grade 3 endocrinopathy that was managed and the participant was asymptomatic; Grade 3 inflammatory reaction attributed to a local antitumor response that resolved to <=Grade 1 within 30 days; concurrent vitiligo or alopecia of any grade; Grade 3 infusion-related reaction that resolved within 6 hours; and any more than or equal to (>=) Grade 3 lymphopenia (unless clinically significant).
Time Frame: From the first dose of study treatment through 28 days after the first dose (up to 28 days)
Population: DLT-evaluable population
Measure: Number; unit: Participant
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Participant | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. TEAEs were events present at baseline that worsened in intensity after administration of study treatment or events absent at baseline that emerged after administration of study treatment.
Time Frame: From study treatment administration (Day 1) to 90 days after the last dose of study treatment or early termination of study (up to 1 year)
Population: As-treated population: all the participants who received any study treatment.
Measure: Number; unit: Participant
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Participant | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1

4. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events
Description: A serious adverse event (SAE) was any AE that resulted in death, immediately life threatening, required (or prolonged) inpatient (or existing) hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly or birth defect in offspring of the participant, or an important medical event that could jeopardize the participant or required medical intervention to prevent one of the outcomes listed above. Treatment-emergent SAEs were defined as SAEs present at baseline that worsened in intensity after administration of study treatment or SAEs absent at baseline that emerged after administration of study treatment.
Time Frame: as for outcome 3
Population: As-treated population
Measure: Number; unit: Participant
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Participant | 4 | 3 | 1 | 5 | 3 | 3 | 3 | 2 | 0

5. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs
Description: Laboratory evaluations of blood and urine samples were performed, including hematology (white blood cell [WBC] count with differential, red blood cell [RBC] count, hematocrit, hemoglobin, platelet count, mean corpuscular volume [MCV], and mean corpuscular hemoglobin concentration [MCHC]); serum chemistry (calcium, chloride, magnesium, creatinine, sodium, blood urea nitrogen [BUN], bicarbonate, glucose, aspartate transaminase [AST], total bilirubin, C-reactive protein, gamma-glutamyl transpeptidase [GGT], lactate dehydrogenase, uric acid, potassium, alanine transaminase [ALT], alkaline phosphatase, albumin, total protein, triglycerides, and cholesterol); urinalysis; and coagulation parameters.
Time Frame: as for outcome 3
Population: As-treated population
Measure: Number; unit: Participant
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Participant
  Anemia | 2 | 2 | 2 | 2 | 2 | 1 | 3 | 1 | 1
  Neutrophil count increased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphopenia | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood iron decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hemoglobin decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutropenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypernatremia | 1 | 1 | 1 | 3 | 2 | 0 | 2 | 0 | 0
  Hypokalemia | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 0
  Aspartate aminotransferase increased | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 1
  Hypomagnesemia | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0
  Blood alkaline phosphatase increased | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
  Hyperglycemia | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
  Blood creatinine increased | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
  Gamma-glutamyltransferase increased | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Hypercalcemia | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hyperkalemia | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
  Hypoalbuminemia | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Hyperuricemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Blood bilirubin increased | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood cholesterol increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Blood glucose increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Blood thyroid stimulating hormone increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypocalcemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypothyroidism | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Iron deficiency | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Liver function test increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Tri-iodothyronine free decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Troponin increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Thyroxine free decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hematuria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Vital Signs and Physical Examination Abnormalities Reported as TEAEs
Description: Vital signs examination included assessment of temperature, blood pressure, pulse rate, and respiratory rate. Physical examination included assessments of head, eyes, ears, nose, throat, respiratory, cardiovascular, gastrointestinal, urogenital, musculoskeletal, neurological, psychiatric, dermatological, hematologic/lymphatic, and endocrine systems. The TEAEs related to these vital sign and physical examination abnormalities were reported.
Time Frame: as for outcome 3
Population: As-treated population
Measure: Number; unit: Participant
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Participant
  Pyrexia | 1 | 2 | 2 | 2 | 0 | 3 | 2 | 0 | 0
  Dyspnea | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 1
  Hypotension | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
  Sinus tachycardia | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Dyspnea exertional | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Tachycardia | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Bradycardia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypertension | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoxia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Wheezing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Reported as TEAEs
Description: Electrocardiogram (ECG) parameters included atrial rate, PR interval, QRS duration, QTC interval, QT interval, and ventricular rate. All 12-lead ECGs performed during the study were obtained in triplicate. The TEAEs related to these ECG evaluation abnormalities were reported.
Time Frame: as for outcome 3
Population: As-treated population
Measure: Number; unit: Participant
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Participant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Best Overall Response (BOR)
Description: Best overall response: Percentage (%) of participants with CR, partial response (PR), stable disease (SD), progressive disease (PD), or non-evaluable disease based on revised Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST v1.1) for monotherapy and combination tremelimumab and durvalumab arms, and Cheson criteria for combination rituximuab arms. Per RECIST v1.1: CR-disappearance of all target/non-target lesions; PR at least a 30% decrease in sum of diameters of target lesions; SD-neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; PD-at least a 20% increase in sum of diameters of target lesions, or a substantial worsening in a non-target lesion, or the appearance of new lesions. Per Cheson criteria: CR-disappearance of all evidence of disease; PR-regression of measurable disease and no new sites; SD-failure to attain CR/PR or PD; PD-any new lesion or increase by at least 50% of previously involved sites from nadir.
Time Frame: From study entry until early termination (up to 1 year)
Population: As-treated population
Measure: Number; unit: Percentage of participants
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Percentage of participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0
  SD | 12.5 | 0 | 33.3 | 28.6 | 33.3 | 14.3 | 0 | 33.3 | 100.0
  PD | 50.0 | 33.3 | 66.7 | 42.9 | 50.0 | 42.9 | 100.0 | 66.7 | 0
  NE | 37.5 | 66.7 | 0 | 28.6 | 0 | 42.9 | 0 | 0 | 0

9. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate was defined as the percentage of participants with confirmed CR or confirmed PR according to revised RECIST v1.1 for monotherapy and combination tremelimumab and durvalumab arms, and Cheson criteria for combination rituximuab arms. Confirmed CR and PR were those that persisted on repeat consecutive assessment >= 4 weeks after the initial documentation of response. Tumor assessments according to revised RECIST v1.1 were defined as follows: CR - disappearance of all target/non-target lesions; PR - at least a 30% decrease in the sum of the diameters of target lesions. Tumor assessments according to Cheson criteria were defined as follows: CR - disappearance of all evidence of disease; PR- regression of measurable disease and no new sites.
Time Frame: From study entry until early termination (up to 1 year)
Population: As-treated population
Measure: Number; unit: Percentage of participants
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Percentage of participants | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0

10. Secondary Outcome: Disease Control Rate
Description: Disease control rate: Percentage of participants with CR, PR, or SD (if they maintained SD for >= 8 weeks) according to revised RECIST v1.1 for monotherapy and combination tremelimumab and durvalumab arms, and Cheson criteria for combination rituximuab arms. Tumor assessments according to revised RECIST v1.1 were defined as follows: CR -disappearance of all target/non-target lesions; PR - at least a 30% decrease in sum of diameters of target lesions; SD - neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; PD - at least a 20% increase in sum of diameters of target lesions, or a substantial worsening in a non-target lesion, or the appearance of new lesions. Tumor assessments according to Cheson criteria were defined as follows: CR- disappearance of all evidence of disease; PR - regression of measurable disease and no new sites; SD- failure to attain CR/PR or PD; PD- any new lesion or increase by at least 50% of previously involved sites from nadir.
Time Frame: From study entry until early termination (up to 1 year)
Population: As-treated population
Measure: Number; unit: Percentage of participants
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Percentage of participants | 12.5 | 0 | 33.3 | 28.6 | 50.0 | 14.3 | 0 | 33.3 | 100.0

11. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was the duration from the first documented objective response to the first documented PD or death due to any cause, whichever occurred first. Progression was based on revised RECIST v1.1 criteria for monotherapy and combination tremelimumab and durvalumab arms, and Cheson criteria for combination rituximuab arms. PD according to revised RECIST v1.1 was defined as: at least a 20% increase in the sum of diameters of target lesions, or a substantial worsening in a non-target lesion, or the appearance of new lesions. PD per Cheson criteria was defined as: any new lesion or increase by at least 50% of previously involved sites from nadir.
Time Frame: From Study entry until early termination (up to 1 year)
Population: All the participants with an OR were included.
Measure: Number; unit: Days
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Days |  |  |  |  | 368 |  |  |  |

12. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was the duration measured from the start of study treatment until the first documentation of PD or death due to any cause, whichever occurred first. Progression was based on revised RECIST v1.1 criteria for monotherapy and combination tremelimumab and durvalumab arms, and Cheson criteria for combination rituximuab arms. PD according to revised RECIST v1.1 was defined as: at least a 20% increase in the sum of diameters of target lesions, or a substantial worsening in a non-target lesion, or the appearance of new lesions. PD per Cheson criteria was defined as: any new lesion or increase by at least 50% of previously involved sites from nadir.
Time Frame: From Study entry until early termination (up to 1 year)
Population: As-treated population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Months | 1.8 [0.9 to 3.5] | 1.8 [1.8 to 1.8] | 1.9 [1.8 to 6.4] | 2.8 [0.7 to 6.7] | 5.6 [1.0 to 17.8] | 1.8 [1.0 to 6.4] | 1.4 [1.0 to 1.8] | 1.0 [0.9 to NA] — Not evaluable due to insufficient number of participants achieved this endpoint | 5.4 [NA to NA] — Not evaluable due to insufficient number of participants achieved this endpoint

13. Secondary Outcome: Overall Survival (OS)
Description: The OS was the duration from the start of study treatment until death due to any cause.
Time Frame: From Study entry until early termination (up to 1 year)
Population: As-treated population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Months | 6.1 [0.9 to NA] — Not evaluable due to insufficient number of participants achieved this endpoint | 6.5 [1.8 to 10.7] | 13.1 [11.2 to NA] — Not evaluable due to insufficient number of participants achieved this endpoint | 6.7 [2.0 to 12.5] | 11.2 [1.2 to 17.8] | NA [1.0 to NA] — Not evaluable due to insufficient number of participants achieved this endpoint | 2.9 [2.5 to NA] — Not evaluable due to insufficient number of participants achieved this endpoint | 3.3 [1.7 to NA] — Not evaluable due to insufficient number of participants achieved this endpoint | NA [NA to NA] — Not evaluable due to insufficient number of participants achieved this endpoint

14. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: The pharmacokinetics (PK) parameter was estimated using the non-compartmental analysis methods, based on the participant serum concentration-time data. The concentration-time curve was the result of blood sampling at specified time points and its measured concentration of MEDI6469
Time Frame: MEDI6469 monotherapy: Days 1, 2, 3, 8, 15, and 29; MEDI6469 + tremelimumab or durvalumab: Days 1, 2, 3, 4, 8, 15, 29, and end of treatment (up to 1 year); MEDI6469 + rituximab: Days 3, 4, 8, 15, 29, 31, 59, every 28 days thereafter, and end of treatment
Population: All the participants who received at least a one dose of MEDI6469 and for whom PK blood samples were collected and evaluated.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
microgram per milliliter | 133.76 (34.87) | 188.87 (59.88) | 49.00 (1.29) | 43.67 (7.99) | 40.21 (8.20) | 42.10 (6.63) | 234.91 (56.05) | 31.68 (5.06) | 289.40 (NA) — Not evaluable due to insufficient number of participants achieved this endpoint

15. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUC0-inf)
Description: The PK parameter was estimated using the non-compartmental analysis methods, based on the participant serum concentration-time data. The concentration-time curve was the result of blood sampling at specified time points and its measured concentration of MEDI6469
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: day*microgram per milliliter
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
day*microgram per milliliter | 556.92 (166.95) | 873.16 (328.74) | 169.34 (18.15) | 183.09 (26.27) | 144.91 (33.07) | 169.65 (45.98) | 998.25 (400.12) | 145.55 (16.86) | 1619.73 (NA) — Not evaluable due to insufficient number of participants achieved this endpoint

16. Secondary Outcome: Systemic Clearance (CL)
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liter per day
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
liter per day | 0.81 (0.224) | 0.84 (0.246) | 1.02 (0.155) | 0.89 (0.132) | 1.04 (0.288) | 1.0 (0.266) | 0.84 (0.173) | 1.11 (0.188) | 0.77 (NA) — Not evaluable due to insufficient number of participants achieved this endpoint

17. Secondary Outcome: Terminal Phase Elimination Half-Life (T1/2)
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Day | 2.83 (0.83) | 3.20 (1.23) | 1.56 (0.04) | 2.86 (0.68) | 2.73 (0.65) | 3.30 (0.68) | 2.98 (1.06) | 3.75 (1.03) | 4.19 (NA) — Not evaluable due to insufficient number of participants achieved this endpoint

18. Secondary Outcome: Number of Participants Positive for Human Anti-mouse Antibodies (HAMA)
Description: The number of participants who developed detectable HAMA are presented. ImmuSTRIP® HAMA IgG ELISA Test System was used for detection, confirmation, and titration of HAMA in human serum with a HAMA positivity cut-off level of 74 nanogram per millilitre (ng/mL).
Time Frame: All treatment arms: Days 8, 15, 29, and end of treatment (up to 1 year). Additionally for MEDI6469 + rituximab arm: Days 3, 31, 59, and every 28 days thereafter until end of treatment (up to 1 year)
Population: All the participants who received at least a one dose of MEDI6469.
Measure: Number; unit: Participant
Arm/Group | MEDI6469 6 mg/kg | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+ Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg + Rituximab 375 mg/m^2
Number analyzed (Participants) | 8 | 6 | 3 | 7 | 6 | 7 | 7 | 3 | 1
Participant | 5 | 4 | 3 | 6 | 5 | 6 | 4 | 1 | 0

ADVERSE EVENTS:
Time Frame: From study treatment administration (Day 1) to 90 days after the last dose of study treatment or early termination of study (up to 1 year)
Arm/Group | MEDI6469 6 Milligram/Kilogram (mg/kg) | MEDI6469 10 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg | MEDI6469 2 mg/kg+Rituximab 375 mg/m^2 | MEDI6469 10 mg/kg+Rituximab 375 mg/m^2
Serious Adverse Events (participants affected / at risk) | 4/8 | 3/6 | 1/3 | 5/7 | 3/6 | 3/7 | 3/7 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 6/8 | 6/6 | 3/3 | 7/7 | 6/6 | 7/7 | 7/7 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI6469 6 Milligram/Kilogram (mg/kg) (N=8) | MEDI6469 10 mg/kg (N=6) | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg (N=3) | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg (N=7) | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg (N=6) | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg (N=7) | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg (N=7) | MEDI6469 2 mg/kg+Rituximab 375 mg/m^2 (N=3) | MEDI6469 10 mg/kg+Rituximab 375 mg/m^2 (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI6469 6 Milligram/Kilogram (mg/kg) (N=8) | MEDI6469 10 mg/kg (N=6) | MEDI6469 2 mg/kg+Tremelimumab 3 mg/kg (N=3) | MEDI6469 2 mg/kg+Tremelimumab 10 mg/kg (N=7) | MEDI6469 2 mg/kg+Durvalumab 3 mg/kg (N=6) | MEDI6469 2 mg/kg+Durvalumab 10 mg/kg (N=7) | MEDI6469 10 mg/kg+Durvalumab 10 mg/kg (N=7) | MEDI6469 2 mg/kg+Rituximab 375 mg/m^2 (N=3) | MEDI6469 10 mg/kg+Rituximab 375 mg/m^2 (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (3) | 2 (3) | 2 (3) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 4 (9) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (3) | 1 (1) | 4 (5) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (5) | 2 (2) | 3 (5) | 4 (6) | 4 (4) | 3 (3) | 3 (4) | 1 (3) | 1 (2)
Influenza like illness (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (4) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 1 (3) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (3) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early at the Sponsor's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.